CLINICAL TRIAL: NCT01151111
Title: Pilot Study of Relaxation Guided Imagery for the Treatment of Motor Fluctuations in Parkinson's Disease's
Brief Title: Relaxation Guided Imagery for Treatment of Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ilana Schlesinger, Director, Movement Disorders Institute, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0457-09-RMB
Record Dates: First submitted 2010-05-18; First posted 2010-06-25 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Relaxation; Visual imagery; Motor fluctuations; Treatment
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Relaxation guided imagery — An individualized relaxation guided imagery session will be conducted. After the session patients will be given a CD with the RGI and asked to listen to it at home.

SUMMARY:
Parkinson's disease patients may have pronounced ON-OFF motor fluctuations. These motor fluctuations are currently treated with medication and surgery, which are limited by their efficacy and side effects. Our study aims to determine whether relaxation guided imagery can alleviate the OFF state of PD patients and therefore can be used as an adjunct to conventional medication.

DETAILED DESCRIPTION:
Parkinson's disease patients with pronounced ON-OFF motor fluctuations without dementia will participate in this study aimed to examine a possible beneficial effect of relaxation guided imagery on motor fluctuations. The study will include a baseline period two sessions of relaxation and a follow-up period. The relaxation sessions will be conducted individually. In one session patients will hear relaxing music and in the second they will undergo relaxation guided imagery. After each relaxation session patients will receive a CD with either relaxing music or RGI to listen to at home. They will be asked to fill out a diary at baseline and after each session. Before and after each relaxation session patients will be examined according to the Unified Parkinson's Disease Rating Scale and the examination will be videotaped. All patients will continue to receive the usual care from their medical providers. The main measure is change in UPDRS and secondary measure is change in daily OFF time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease suffering from motor fluctuations
* H&Y >2

Exclusion Criteria:

* Dementia
* hearing impairment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Unified Parkinson's Disease Rating Scale (UPDRS) | 30 minutes
  * Unified Parkinson's Disease Rating Scale (UPDRS) score after RGI as compared to baseline
  * OFF time after RGI as compared to baseline

SECONDARY OUTCOMES:
Change from baseline to week 2 in Clinical Global Impression Scale (CGI) | 2 weeks
  Patient will fill out a CGI
Change from baseline to week 2 in PDQ39 | 2 weeks
  PDQ39 questionaire will be filled out by the patient
Change from baseline to minutes 30 of Unified Parkinson's Disease Rating Scale (UPDRS) after relaxing music | 30 minutes
  * Unified Parkinson's Disease Rating Scale (UPDRS) score after relaxing music as compared to baseline
  * OFF time after relaxing music as compared to baseline
Change from baseline to week 2 in the number of OFF hours | 2 weeks
  The mean number of daily OFF hours over 3 days after visit.
Change from baseline to month 3 in PDQ39 | 3 months
  PDQ39 questionaire will be filled out by the patient
Change from baseline to month 3 in Clinical Global Impression Scale (CGI) | 3 months
  Patient will fill out a CGI
Change from baseline to week 1 in the number of OFF hours | 1 week
  The mean number of daily OFF hours over 3 days after visit

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Schlesinger, M.D., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Ilana Schleainger, Haifa, Israel